CLINICAL TRIAL: NCT02174731
Title: A Phase 3, Multicenter, Randomized, Open-label, Active-Controlled Study of the Safety and Efficacy of Roxadustat in the Treatment of Anemia in Dialysis Patients
Brief Title: Safety and Efficacy Study of Roxadustat to Treat Anemia in Patients With Chronic Kidney Disease, on Dialysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5740C00002
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Anemia
Keywords: Renal,; CKD,; Epoetin alfa,; Roxadustat,; dialysis,; anemia
MeSH Terms: conditions — Anemia | interventions — roxadustat; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental)
  Interventions: Drug: Roxadustat
- Epoetin alfa (Active Comparator)
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be administered orally three times a week (TIW) to achieve an Hb level of 11 g/dL and maintain a Hb level of 11±1 g/dL.
  Arms: Roxadustat
Drug: Epoetin alfa — Epoetin alfa will be administered TIW consistent with approved prescribing information for epoetin alfa to achieve an Hb level of 11 g/dL and maintain a Hb level of 11±1 g/dL.
  Arms: Epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of roxadustat compared to epoetin alfa for the treatment of anemia in chronic kidney disease patients on dialysis.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, open-label, active-controlled study to evaluate the efficacy and safety of roxadustat compared to epoetin alfa for the treatment of anemia in dialysis patients. Patients on hemodialysis (HD) or peritoneal dialysis (PD) who have been treated with an erythropoietin analogue or have an indication for treatment with an erythropoietin analogue will be evaluated for eligibility and randomized at a 1:1 ratio to treatment with roxadustat (with discontinuation of prior erythropoietin analogue therapy) or to an active-control group treated with epoetin alfa

ELIGIBILITY:
Inclusion criteria:

1. Provision of Informed Consent prior to any study specific procedures
2. Age ≥18 years at screening visit 1
3. Previous versions of the protocol prior to US amendment ver 6.0 and outside of US amendment ver 7.0:

   Receiving or initiating hemodialysis or peritoneal dialysis for treatment of native kidney end-stage renal disease (ESRD) at least 30 days prior to visit 1. Patients treated with hemodialysis must have access consisting of an arteriovenous fistula, AV graft, or tunneled (permanent) catheter. Patients on peritoneal dialysis must have a functioning peritoneal dialysis catheter in place.

   Starting with US amendment ver. 6.0 and outside of US amendment ver 7.0 (changed to recruit incident dialysis patients only):

   Receiving or initiating hemodialysis or peritoneal dialysis for treatment of native kidney end-stage renal disease (ESRD) for a minimum of 2 weeks and a maximum of 4 months prior to randomization. Patients treated with hemodialysis must have access consisting of an arteriovenous fistula, AV graft, or tunneled (permanent) catheter. Patients on peritoneal dialysis must have a functioning peritoneal dialysis catheter in place.
4. Two central laboratory Hb values during the screening period, obtained at least 7 days apart, must be <12 g/dL in patients currently treated with an erythropoietin analogue or <10 g/dL in patients not currently treated with an erythropoietin analogue. Patients are considered not currently treated if they have not received either Mircera® for at least 8 weeks or any other erythropoietin analogue for at least 4 weeks prior to visit 1.
5. Ferritin ≥100 ng/mL at randomization (obtained from screening visit)
6. TSAT ≥20% at randomization (obtained from screening visit)
7. Serum folate level ≥ lower limit of normal (LLN) at randomization (obtained from screening visit)
8. Serum vitamin B12 level ≥ LLN at randomization (obtained from screening visit)
9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3x upper limit of normal (ULN), and total bilirubin (Tbili) ≤1.5 x ULN at randomization (obtained from screening visit)
10. Body weight 45 to 160 kg (prescribed dry weight)

Exclusion criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous randomisation in the present study
3. New York Heart Association Class III or IV congestive heart failure at enrolment
4. Myocardial infarction, acute coronary syndrome, stroke, seizure or a thrombotic/thromboembolic event (e.g., deep vein thrombosis or pulmonary embolism) within 12 weeks prior to randomization
5. History of chronic liver disease (e.g., chronic infectious hepatitis, chronic auto-immune liver disease, cirrhosis or fibrosis of the liver)
6. Known hereditary hematologic disease such as thalassemia, sickle cell anemia, a history of pure red cell aplasia or other known causes for anemia other than CKD
7. Known and untreated retinal vein occlusion or known and untreated proliferative diabetic retinopathy (risk for retinal vein thrombosis)
8. Diagnosis or suspicion (e.g. complex kidney cyst of Bosniak Category IIF, III or IV) of renal cell carcinoma on renal ultrasound (or other imaging procedure e.g. CT scan or MRI) conducted at screening or within 12 weeks prior to randomization.
9. Uncontrolled hypertension at the time of randomization (defined as systolic BP ≥180 mmHg or diastolic BP ≥100 mmHg on repeated measurement post-dialysis in hemodialysis patients or at any time in peritoneal dialysis patients), contraindication to epoetin alfa treatment (e.g., pure red cell aplasia, hypersensitivity or know inability to tolerate epoetin alfa)
10. History of prostate cancer, breast cancer or any other malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ or resected colonic polyps.
11. Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus antibody (anti-HCV Ab)
12. Chronic inflammatory diseases such as rheumatoid arthritis, SLE, ankylosing spondylitis, psoriatic arthritis or inflammatory bowel disease that is determined to be the principal cause of anemia
13. Known hemosiderosis, hemochromatosis or hypercoagulable condition
14. Any prior organ transplant with the exception of an autologous renal transplant or a renal transplant that was subsequently removed ("explanted") or scheduled organ transplantation date
15. Any red blood cell (RBC) transfusion during the screening period
16. Any current condition leading to active significant blood loss
17. Any prior treatment with roxadustat or a hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI)
18. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within the month preceding the first administration of IP in this study. (Note: patients consented and screened, but not randomized in this study or a previous study are not excluded)
19. History of alcohol or drug abuse within 2 years prior to randomization
20. Females of childbearing potential, unless using contraception as detailed in the protocol or sexual abstinence (see Section 3.8)
21. Pregnant or breastfeeding females
22. Known allergy to the investigational product or any of its ingredients
23. Any medical condition, including active, clinically significant infection, that in the opinion of the investigator or Sponsor may pose a safety risk to a patient in this study, which may confound efficacy or safety assessment, or may interfere with study participation

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2133 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Principal Investigator — Chief Division of Kidney Diseases and Hypertension, North Shore University Hospital, Great Neck, NY, USA; Mark Houser, MD, Study Director — AZ R&D, Gaithersburg, USA
Locations (160):
- United States (44):
  - Research Site, Huntsville, Alabama
  - Research Site, El Centro, California
  - Research Site, Fairfield, California
  - Research Site, Glendale, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Northridge, California
  - Research Site, Ontario, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, Sun Valley, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Miami Gardens, Florida
  - Research Site, River Forest, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lanham, Maryland
  - Research Site, Plymouth, Massachusetts
  - Research Site, Roseville, Michigan
  - Research Site, Gulfport, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Paterson, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Orchard Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Shawnee, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Newport News, Virginia
  - Research Site, Sterling, Virginia
  - Research Site, Bluefield, West Virginia
- Australia (7):
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, Launceston
  - Research Site, Prahan
  - Research Site, St Leonards
  - Research Site, Wahroonga
- Bulgaria (12):
  - Research Site, Botevgrad
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Haskovo
  - Research Site, Razlog
  - Research Site, Samokov
  - Research Site, Sandanski
  - Research Site, Shumen
  - Research Site, Silistra
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Yambol
- Canada (11):
  - Research Site, Edmonton, Alberta
  - Research Site, Kamloops, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, Sydney, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (6):
  - Research Site, Brno
  - Research Site, Prague
  - Research Site, Rychnov nad Kněžnou
  - Research Site, Slaný
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Hungary (7):
  - Research Site, Ajka
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
- India (13):
  - Research Site, Chennai
  - Research Site, Ghaziabad NCR
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Maharashtra
  - Research Site, Mumbai
  - Research Site, Mysore
  - Research Site, Nadiād
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vellore
  - Research Site, Vijayawada
- Mexico (4):
  - Research Site, Aguascalientes
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Veracruz
- Research Site, Lima, Peru
- Philippines (2):
  - Research Site, Cebu City
  - Research Site, Iloilo City
- Poland (8):
  - Research Site, Ciechanów
  - Research Site, Gmina Końskie
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Pszczyna
  - Research Site, Suwałki
  - Research Site, Tarnów
  - Research Site, Warsaw
- Russia (13):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Kráľovský Chlmec
  - Research Site, Nové Zámky
  - Research Site, Zvolen
- Spain (7):
  - Research Site, Almería
  - Research Site, Barcelona
  - Research Site, Granollers (Barcelona)
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Tarragona
  - Research Site, Valencia
- Sweden (4):
  - Research Site, Karlstad
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Västerås
- Research Site, Bangkok, Thailand
- Ukraine (10):
  - Research Site, Chernivtsi
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- Vietnam (4):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Hochiminh
  - Research Site, Huế

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Martin S, Jiletcovici A, Dellanna F, Akizawa T, Barratt J. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Four Global Roxadustat Phase 3 Trials. Adv Ther. 2024 Apr;41(4):1553-1575. doi: 10.1007/s12325-023-02728-2. Epub 2024 Feb 16. PMID 38363466
- [Derived] Barratt J, Dellanna F, Portoles J, Choukroun G, De Nicola L, Young J, Dimkovic N, Reusch M. Safety of Roxadustat Versus Erythropoiesis-Stimulating Agents in Patients with Anemia of Non-dialysis-Dependent or Incident-to-Dialysis Chronic Kidney Disease: Pooled Analysis of Four Phase 3 Studies. Adv Ther. 2023 Apr;40(4):1546-1559. doi: 10.1007/s12325-023-02433-0. Epub 2023 Feb 7. PMID 36749544
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Fishbane S, Pollock CA, El-Shahawy M, Escudero ET, Rastogi A, Van BP, Frison L, Houser M, Pola M, Little DJ, Guzman N, Pergola PE. Roxadustat Versus Epoetin Alfa for Treating Anemia in Patients with Chronic Kidney Disease on Dialysis: Results from the Randomized Phase 3 ROCKIES Study. J Am Soc Nephrol. 2022 Apr;33(4):850-866. doi: 10.1681/ASN.2020111638. PMID 35361724
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5740C00002&attachmentIdentifier=1cab3812-b878-4cc4-9c31-d56a8992967c&fileName=D5740C00002_redacted_CSP_from_PRS.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5740C00002&attachmentIdentifier=4c981c0f-6734-4567-b362-92b2e86d7fdf&fileName=D5740C00002-SAP-ed4_Redacted_(1).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 197 centers in 18 countries worldwide across the United States (US), Canada, Latin America, Australia, Asia and Europe between 01 July 2014 and 26 September 2018. Participants with chronic kidney disease (CKD) who were on dialysis were recruited in this study.
Pre-assignment Details: Study had a screening period (up to 6 weeks), treatment period (up to 4 years) and follow-up period (4 weeks after treatment period for those who completed treatment). 2133 participants were randomized, of which 2106 were included in the analysis and 27 were excluded. Only participants included in the analysis are presented in the participant flow.
Groups:
- Roxadustat: Participants received roxadustat tablets orally three times a week (TIW) throughout the treatment period (up to 4 years). For hemodialysis (HD) participants, it was recommended that roxadustat was taken after completion of the HD session. For participants treated with an erythropoietin analogue at study entry, selection of initial roxadustat dose was based on the participant's erythropoietin analogue dose at screening Visit 1. Participants not treated with an erythropoietin analogue at study entry initiated roxadustat using a tiered, weight-based dosing scheme. Doses were titrated to achieve and maintain hemoglobin (Hb) values of 11±1 grams per deciliter (g/dL). Dose adjustments were permitted starting at Week 4 and at intervals of every 4 weeks using a dose adjustment algorithm.
- Epoetin Alfa: Participants received epoetin alfa (only use of Procrit®, Eprex® and Epogen® permitted in the study) subcutaneous (SC) or intravenous (IV) injection TIW, except for participants treated with epoetin alfa in a less frequent regimen prior to study entry. For participants treated with an erythropoietin analogue at study entry, the initial dose of epoetin alfa was the actual dose administered at screening Visit 1. Participants treated with darbepoetin alfa or methoxy polyethylene glycol-epoetin beta prior to study entry initially received epoetin alfa at doses based on a conversion factor. For participants not treated with an erythropoietin analogue at study entry, the initial dose of epoetin alfa was 50 international unit per kilogram (IU/kg) TIW. Dose adjustments were to be consistent with local approved prescribing information.
Period: Overall Study
Arm/Group | Roxadustat | Epoetin Alfa
Started (Randomized and included in the analysis) | 1051 | 1055
Received Treatment | 1048 | 1053
Completed (Completed the study) | 982 | 990
Not Completed | 69 | 65
Not completed — Participant decision | 67 | 64
Not completed — Incorrect enrolment before randomization | 0 | 1
Not completed — Missing | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat (ITT) analysis set included all participants who were randomized to investigational product (IP) irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis.
Groups:
- Roxadustat: Participants received roxadustat tablets orally TIW throughout the treatment period (up to 4 years). For HD participants, it was recommended that roxadustat was taken after completion of the HD session. For participants treated with an erythropoietin analogue at study entry, selection of initial roxadustat dose was based on the participant's erythropoietin analogue dose at screening Visit 1. Participants not treated with an erythropoietin analogue at study entry initiated roxadustat using a tiered, weight-based dosing scheme. Doses were titrated to achieve and maintain Hb values of 11±1 g/dL. Dose adjustments were permitted starting at Week 4 and at intervals of every 4 weeks using a dose adjustment algorithm.
- Epoetin Alfa: Participants received epoetin alfa (only use of Procrit®, Eprex® and Epogen® permitted in the study) SC or IV injection TIW, except for participants treated with epoetin alfa in a less frequent regimen prior to study entry. For participants treated with an erythropoietin analogue at study entry, the initial dose of epoetin alfa was the actual dose administered at screening Visit 1. Participants treated with darbepoetin alfa or methoxy polyethylene glycol-epoetin beta prior to study entry initially received epoetin alfa at doses based on a conversion factor. For participants not treated with an erythropoietin analogue at study entry, the initial dose of epoetin alfa was 50 IU/kg TIW. Dose adjustments were to be consistent with local approved prescribing information.
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Epoetin Alfa | Total
Number analyzed (Participants) | 1051 | 1055 | 2106
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (15.30) | 54.5 (14.97) | 54.0 (15.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 426 | 429 | 855
  Male | 625 | 626 | 1251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 268 | 271 | 539
  Not Hispanic or Latino | 783 | 784 | 1567
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 597 | 598 | 1195
  Black of African American | 148 | 158 | 306
  Asian | 208 | 198 | 406
  Native Hawaiian or other Pacific Islander | 5 | 3 | 8
  American Indian or Alaska Native | 50 | 62 | 112
  Other | 43 | 36 | 79

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hb Averaged Over Week 28 to Week 52
Description: Baseline Hb was defined as the mean of the three last central laboratory Hb values from the screening and randomization visits. Mean change in Hb from baseline to the participants mean level from Week 28 to Week 52 was analyzed using a missing at random (MAR) based multiple imputation Analysis of Covariance (ANCOVA). Baseline Hb was used as a covariate and treatment group, cardiovascular (CV) history, geographic region and dialysis duration as fixed effects. The adjusted least squares (LS) mean estimates of change from baseline during Week 28 to Week 52 are presented.
Time Frame: Baseline (Day 1, Week 0), Week 28 to 52
Population: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 1003 | 1016
g/dL | 0.77 (0.041) | 0.68 (0.040)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority of roxadustat versus epoetin alfa was declared if the lower bound of the 95% confidence interval (CI) of the difference between roxadustat and epoetin alfa exceeded -0.75. Non-inferiority p-value is 1-sided; p < 0.001, ANCOVA; Least Square Mean Difference = 0.09, 95% CI 2-sided [0.01 to 0.18], Standard Error of Mean 0.044 — Difference between groups (roxadustat minus Epoetin alfa) in LS mean changes

2. Secondary Outcome: Change in Hb From Baseline to the Mean Level During the Evaluation Period (Week 28 to Week 36) Without Having Received Rescue Therapy Within 6 Weeks Prior to and During the 8-Week Evaluation Period
Description: Baseline Hb was defined as the mean of the three last central laboratory Hb values from the screening and randomization visits. Mean change in Hb from baseline to the participants mean level from Week 28 to Week 36,without having received rescue therapy within 6 weeks prior to and during this 8 week evaluation period was analysed using Mixed Model of Repeated Measures (MMRM). Baseline Hb was used as a covariate and treatment group, CV history, geographic region and dialysis duration as fixed effects. The adjusted LS mean estimates of change from baseline during Week 28 to Week 36 are presented for participants that did not receive rescue therapy within 6 weeks prior to and during this 8-week evaluation period.
Time Frame: Baseline (Day 1, Week 0), Week 28 to 36
Population: The Per Protocol Set (PPS) included all randomized participants without important protocol deviations who had received at least 8 weeks of study treatment and had valid corresponding Hb measurements. Participants from the PPS, with data available for analysis are presented.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 836 | 864
g/dL | 0.88 (0.044) | 0.74 (0.043)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority of roxadustat versus epoetin alfa was declared if the lower bound of the 95% CI of the difference between roxadustat and epoetin alfa exceeded -0.75. Non-inferiority p-value is 1-sided; p < 0.001, MMRM; Least Square Mean Difference = 0.14, 95% CI 2-sided [0.03 to 0.25], Standard Error of Mean 0.056 — Difference between groups (roxadustat minus Epoetin alfa) in LS mean change

3. Secondary Outcome: Proportion of Total Time of Hb Within the Interval of >=10 g/dL From Week 28 to Week 52
Description: The proportion of total time was computed as follows: For each participant, the recorded Hb values were first linearly interpolated between measurements. The time this interpolated curve was >=10 g/dL was computed and subsequently divided by the time between the measurements from Week 28 to Week 52. The difference between roxadustat and epoetin alfa were compared using ANCOVA. Baseline Hb was used as a covariate and the treatment groups, CV history, geographic region and dialysis duration as fixed effects.
Time Frame: Week 28 to 52
Population: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis. Participants without any Hb measurements from Week 28 were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: proportion of total time
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 896 | 941
proportion of total time | 0.79 (0.012) | 0.76 (0.012)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority of roxadustat versus epoetin alfa was declared if the lower bound of the 95% CI of the difference between roxadustat and epoetin alfa exceeded -0.15. Non-inferiority p-value is 1-sided; p < 0.001, ANCOVA; Least Square Mean Difference = 0.03, 95% CI 2-sided [0.00 to 0.05], Standard Error of Mean 0.013 — Difference between groups (roxadustat minus Epoetin alfa) in LS mean

4. Secondary Outcome: Proportion of Total Time of Hb Within the Interval of 10 to 12 g/dL From Week 28 to Week 52
Description: The proportion of total time was computed as follows: For each participant, the recorded Hb values were first linearly interpolated between measurements. The time this interpolated curve was within 10-12 g/dL was computed and subsequently divided by the time between the measurement from Week 28 to 52. The difference between roxadustat and epoetin alfa were compared using ANCOVA. Baseline Hb was used as a covariate and the treatment groups, CV history, geographic region and dialysis duration as fixed effects.
Time Frame: Week 28 to 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: proportion of total time
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 896 | 941
proportion of total time | 0.65 (0.013) | 0.63 (0.012)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < 0.001, ANCOVA; Least Square Mean Difference = 0.02, 95% CI 2-sided [-0.01 to 0.05], Standard Error of Mean 0.014 — Difference between groups (roxadustat minus Epoetin alfa) in LS mean

5. Secondary Outcome: Mean Change in Low-Density Lipoprotein (LDL) Cholesterol From Baseline to Week 24
Description: Baseline LDL was defined as the last result obtained prior to randomization. Mean changes in LDL cholesterol from baseline to Week 24 was analysed using ANCOVA. Baseline Hb and baseline LDL were used as covariates and treatment groups, CV history, geographic region and dialysis duration as fixed effects. The adjusted LS mean estimates of change from baseline to Week 24 are presented.
Time Frame: Baseline (Day 1, Week 0) to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimole per liter
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 902 | 937
millimole per liter | -0.38 (0.026) | -0.05 (0.026)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Superiority — Superiority was also declared as the lower bound of the 95% CI exceeded 0 and p-value was lower than 0.05; p < 0.001, ANCOVA; Least Square Mean Difference = -0.33, 95% CI 2-sided [-0.39 to -0.27], Standard Error of Mean 0.030 — Difference between groups (roxadustat minus Epoetin alfa) in LS mean

6. Secondary Outcome: Mean Change in Hb From Baseline to the Participant's Mean Level Between Week 28 to Week 52 in Participants With Baseline High-Sensitivity C-Reactive Protein (hsCRP) Greater Than the Upper Limit of Normal (ULN)
Description: Baseline hsCRP was quantified from stored biomarker samples obtained at randomization. Baseline Hb is defined as the mean of the three last central laboratory Hb values from the screening and randomization visits. Changes in Hb from baseline to mean value during Weeks 28 to 52 in participants with baseline hsCRP >ULN was analyzed using a MAR based multiple imputation ANCOVA. Baseline Hb was used as a covariate and treatment group, CV history, geographic region and dialysis duration as fixed effects. The adjusted LS mean estimates of change from baseline during Week 28 to Week 52 are presented.
Time Frame: Baseline (Day 1, Week 0), Week 28 to 52
Population: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis. Only participants who consented to the use of donated biomarker samples and had baseline hsCRP >ULN were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 280 | 301
g/dL | 0.80 (0.077) | 0.59 (0.076)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.001, ANCOVA; MAR-based multiple imputation; Least Square Mean Difference = 0.20, 95% CI 2-sided [0.04 to 0.36], Standard Error of Mean 0.081 — Difference between groups (roxadustat minus Epoetin alfa) in LS mean

7. Secondary Outcome: Mean Monthly IV Iron Use From Week 36 to End of Study (EOS)
Description: Oral iron supplementation was allowed for both treatment groups without restriction. Oral iron was recommended for dietary supplementation to support erythropoiesis and as the first line treatment for prevention and treatment of iron deficiency, unless the participant was intolerant to this route of treatment. In participants receiving roxadustat, the Investigator was allowed to initiate the use of an approved IV iron supplement if a participant's Hb value had not sufficiently responded to 2 or more dose increases of the IP, and ferritin <100 nanogram per milliliter (ng/mL) or transferrin saturation (TSAT) <20%. IP treatment was allowed to continue during IV iron administration. Discontinuation of IV iron supplementation was recommended once the participant was no longer considered to be iron deficient (ferritin >100 ng/mL and TSAT >20%).
Time Frame: Week 36 to EOS (4 weeks after the treatment period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per month
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 885 | 920
milligram per month | 58.71 (236.12) | 91.37 (225.64)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Superiority; p < 0.0001, Wilcoxon Rank Sum Test

8. Secondary Outcome: Time-To-First Administration of RBC Transfusion as Rescue Therapy
Description: Time-to-first RBC transfusion as rescue therapy was calculated as (date of first occurrence of any RBC transfusion as rescue therapy, or date of censoring if no event had occurred) - (date of first dose of IP) + 1. Event rate was calculated as (number of participants with event) divided by (the total number of days at risk for event across all participants in given group divided by 365.25) multiplied by 100. The event rate is presented for participants with events.
Time Frame: Baseline (Day 1, Week 0) up to EOS (4 weeks after the treatment period)
Population: The on-treatment+3 days safety analysis set included all participants who received at least 1 dose of randomized IP, except for those excluded from analysis. Participants were censored at 3 days after the last administration of the IP.
Measure: Number; unit: events per 100 participant years
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 1048 | 1053
events per 100 participant years | 6.0 | 7.2
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Test type: Non-Inferiority — Non-inferiority of roxadustat versus epoetin alfa was declared if the upper bound of the HR 95% CI of the difference between roxadustat and epoetin alfa was less than or equal to 1.8. Non-inferiority p-value is 1-sided. The CIs were from Wald and ties were calculated using the Efron method; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.64 to 1.07]

ADVERSE EVENTS:
Time Frame: From the first dose of IP administration (Day 1, Week 0) to 28 days after the last administration of the IP, with treatment duration up to 4 years.
Description: The on-treatment+28 days safety analysis set included all participants who received at least 1 dose of randomized IP, except for those excluded from analysis. Participants were censored at 28 days after the last administration of the IP. All-Cause Mortality represents all deaths due to any cause.
Arm/Group | Roxadustat | Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 247/1048 | 231/1053
Serious Adverse Events (participants affected / at risk) | 604/1048 | 606/1053
Other Adverse Events (participants affected / at risk) | 391/1048 | 360/1053
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=1048) | Epoetin Alfa (N=1053)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone marrow reticulin fibrosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 6 (6) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 39 (49) | 41 (46)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (12) | 18 (21)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 10 (11) | 5 (5)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 24 (35) | 29 (43)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 2 (2)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 17 (17) | 16 (18)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 14 (15) | 6 (6)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 6 (6)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis uraemic (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 2 (2)
Right ventricular failure (Cardiac disorders) | 0 (0) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 5 (6) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 3 (3) | 2 (2)
Hyperparathyroidism tertiary (Endocrine disorders) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (8)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (5) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 4 (5)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 5 (6) | 4 (5)
Catheter site haemorrhage (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 3 (3) | 3 (3)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 2 (2)
Dialysis membrane reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 3 (3)
Arteriovenous fistula site infection (Infections and infestations) | 6 (6) | 3 (3)
Arthritis bacterial (Infections and infestations) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 4 (5) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 2 (2)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 12 (13) | 16 (18)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 3 (4)
Cystitis (Infections and infestations) | 5 (5) | 0 (0)
Device related infection (Infections and infestations) | 11 (12) | 11 (15)
Device related sepsis (Infections and infestations) | 5 (5) | 7 (8)
Diabetic foot infection (Infections and infestations) | 3 (3) | 2 (2)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 9 (10) | 11 (13)
Gas gangrene (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 11 (13) | 6 (6)
Gastroenteritis aeromonas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 2 (2) | 1 (1)
Hiv infection (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis c (Infections and infestations) | 1 (1) | 1 (1)
Implant site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Infected fistula (Infections and infestations) | 2 (2) | 1 (1)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (3)
Influenza (Infections and infestations) | 5 (6) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (3)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Neurocysticercosis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 10 (17) | 10 (10)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 24 (28) | 24 (37)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 70 (80) | 78 (92)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (3) | 2 (2)
Pyelonephritis chronic (Infections and infestations) | 3 (4) | 1 (1)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (2)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 40 (44) | 40 (46)
Septic shock (Infections and infestations) | 12 (13) | 13 (15)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Tetanus (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 2 (2)
Tuberculosis (Infections and infestations) | 0 (0) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (2)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 6 (13) | 10 (13)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Kidney rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Post procedural urine leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 16 (20) | 13 (15)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Stress echocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Synovial fluid crystal present (Investigations) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 7 (10) | 3 (7)
Fluid retention (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
5q minus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain hypoxia (Nervous system disorders) | 2 (2) | 0 (0)
Brain injury (Nervous system disorders) | 3 (3) | 0 (0)
Brain oedema (Nervous system disorders) | 4 (4) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 14 (14) | 12 (12)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 8 (8) | 6 (6)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 4 (4) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 10 (10) | 11 (12)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 (2) | 1 (1)
Postresuscitation encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Sciatic nerve neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 5 (6) | 11 (13)
Tardive dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Tonic convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo cns origin (Nervous system disorders) | 0 (0) | 1 (1)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 5 (7) | 3 (3)
Device occlusion (Product Issues) | 2 (2) | 0 (0)
Thrombosis in device (Product Issues) | 3 (3) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Illusion (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 6 (6) | 6 (6)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 13 (15) | 11 (12)
End stage renal disease (Renal and urinary disorders) | 5 (5) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (11)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 9 (10)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 7 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 20 (22)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (7)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 4 (7) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (2) | 0 (0)
Brachiocephalic vein occlusion (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 11 (11) | 0 (0)
Diabetic microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 3 (5)
Hypertension (Vascular disorders) | 12 (16) | 12 (13)
Hypertensive crisis (Vascular disorders) | 24 (32) | 36 (38)
Hypertensive emergency (Vascular disorders) | 24 (26) | 31 (33)
Hypotension (Vascular disorders) | 17 (18) | 18 (20)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 3 (3) | 2 (3)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 4 (5) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 2 (4) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 5 (7) | 5 (5)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 3 (3)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Superior vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous stenosis (Vascular disorders) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 8 (13) | 8 (8)
Angina unstable (Cardiac disorders) | 5 (8) | 6 (6)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (4) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 6 (6) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 7 (7)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 13 (14) | 10 (10)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 7 (7) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 4 (4)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 4 (5)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 2 (3)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 3 (3)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (15) | 10 (10)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal wall mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 11 (15) | 5 (5)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 (24) | 21 (25)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 5 (10) | 4 (4)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal metaplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Malabsorption (Gastrointestinal disorders) | 1 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 5 (6)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 8 (9)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8) | 9 (13)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 4 (4)
Complication associated with device (General disorders) | 0 (0) | 2 (2)
Complication of device insertion (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 21 (21) | 23 (23)
Device related thrombosis (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Haemorrhagic cyst (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 4 (4)
Non-cardiac chest pain (General disorders) | 12 (15) | 9 (11)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 8 (10)
Sudden death (General disorders) | 6 (6) | 5 (5)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (3)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 6 (6)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (5) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 1 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 2 (2)
Transplant rejection (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Abscess of salivary gland (Infections and infestations) | 0 (0) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1)
Acute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 2 (2) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacterial colitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 3 (3) | 1 (1)
Balanoposthitis infective (Infections and infestations) | 1 (1) | 0 (0)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (7) | 5 (5)
Campylobacter colitis (Infections and infestations) | 0 (0) | 1 (1)
Candida pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Catheter site abscess (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 3 (4) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 3 (3)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 5 (5) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (3)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (3) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2)
Joint abscess (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 2 (2)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium abscessus infection (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 3 (3)
Renal cyst infection (Infections and infestations) | 0 (0) | 1 (3)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 7 (7)
Septic embolus (Infections and infestations) | 2 (2) | 1 (1)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 3 (4) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 4 (4) | 3 (3)
Systemic viral infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 13 (13)
Urosepsis (Infections and infestations) | 2 (2) | 3 (3)
Vascular access site infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 3 (3)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 9 (10) | 5 (6)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 37 (46) | 31 (35)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 6 (8)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 4 (5) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve root injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Echocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Human rhinovirus test positive (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pulse absent (Investigations) | 1 (1) | 0 (0)
Respirovirus test positive (Investigations) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 32 (55) | 29 (35)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (10) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 27 (32) | 21 (26)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 19 (22) | 11 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Calcification of muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 3 (3) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 5 (5) | 4 (4)
Cognitive disorder (Nervous system disorders) | 1 (2) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 4 (4)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 5 (5) | 3 (3)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 13 (14) | 7 (7)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 10 (13) | 6 (6)
Device dislocation (Product Issues) | 5 (6) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 7 (7) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 14 (19)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (9)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 6 (7) | 6 (8)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic vein stenosis (Vascular disorders) | 1 (1) | 1 (1)
Brachiocephalic vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 2 (2) | 3 (3)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 2 (2)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 3 (5)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 2 (3)
Peripheral vascular disorder (Vascular disorders) | 5 (5) | 6 (6)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 4 (4) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Vascular compression (Vascular disorders) | 0 (0) | 1 (1)
Venous aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=1048) | Epoetin Alfa (N=1053)
Diarrhoea (Gastrointestinal disorders) | 114 (159) | 101 (153)
Nausea (Gastrointestinal disorders) | 61 (72) | 65 (94)
Vomiting (Gastrointestinal disorders) | 60 (69) | 52 (64)
Bronchitis (Infections and infestations) | 43 (67) | 61 (95)
Upper respiratory tract infection (Infections and infestations) | 70 (102) | 54 (77)
Headache (Nervous system disorders) | 79 (91) | 56 (85)
Cough (Respiratory, thoracic and mediastinal disorders) | 61 (77) | 62 (76)
Hypertension (Vascular disorders) | 85 (130) | 85 (124)
Hypotension (Vascular disorders) | 64 (79) | 54 (83)

LIMITATIONS AND CAVEATS:
27 participants were excluded from the analysis due to Good Clinical Practice violations or system technical issues (17 in the roxadustat group and 10 in the epoetin alfa group).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02174731/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02174731/SAP_001.pdf